CLINICAL TRIAL: NCT03105076
Title: Impact of Decision Aids on Breast Cancer Surgery Choice: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Principal Investigator, Ka-Wai Tam, Director of Shared Decision Making Resource Center, Taipei Medical University Shuang Ho Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: W105HHC-07
Record Dates: First submitted 2017-03-29; First posted 2017-04-07 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Decision Support Techniques

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DAs group (Experimental): Shared decision making using decision aids
  Interventions: Other: Decision aids
- Control group (No Intervention): Standard oral explanation guided with booklets

INTERVENTIONS:
Other: Decision aids — Shared decision making with decision aids
  Arms: DAs group

SUMMARY:
Both simple mastectomy and breast conservation therapy (BCT) with radiotherapy yield similar survival rates in breast cancer. These two treatment strategies have diverted cosmetic outcome and convenience. Thus, shared decision making (SDM) is necessary to aid patients to choose an appropriate treatment that suits thier needs. We have developed a decision aids (DAs) and plan to conduct a randomized controlled trial (RCT) to evaluate its impact on cancer patients. The measurements include a battery of interview-based questionnaires and evaluations of decision regret and postsurgical depression. We expect the DAs would benefit the intervention group in the aspects of knowledge, communication and anxiety status during and after thier treatment sessions.

DETAILED DESCRIPTION:
Background:

For women with early-stage breast cancer, both simple mastectomy and breast conservation therapy (BCT) with radiotherapy yield similar survival rates, making psychological adjustment and quality-of-life issues pivotal in treatment choice. Using decision aids (DAs) is one way to provide information to patients and to involve them in making decisions about their treatment. We have developed a DAs to be administered after consultation for Taiwanese women deciding on breast surgery, and plan to conduct a randomized controlled trial (RCT) to evaluate the benefit of DAs on breast surgery decision making.

Patients and Methods:

Decision aids are interventions designed to help patients with early breast cancer to make deliberate choices among treatment options by providing information on those options and any potential outcome relevant to different breast cancer surgeries. Women considering breast cancer surgery are randomly assigned to receive a DAs or the standard oral conversation (control condition) after initial consultation, wherein surgeons disclosed the diagnosis and discussed treatment options with patients. Participants complete interview-based questionnaires 1 day before and 4 weeks after surgery. Primary outcome measures 1 day before surgery are decisional conflict and decision-making difficulties after consultation. Secondary outcomes are decision regret and postsurgical depression 1 month after surgery.

Hypothesis:

The DAs group are predicted to lower decisional conflict scores before surgery, and lower decision regret scores and depression scores 1 month after surgery compared with women in the control arm. Our study hopes to support the efficacy of DAs in helping breast cancer women to arrive at their breast surgery decision.

ELIGIBILITY:
Inclusion Criteria:

* Taiwanese women newly diagnosed with stage 0 to 3 breast cancer (including patients with ductal carcinoma in situ), who were suitable for breast surgery
* Patients who were able to give consent and complete the interview

Exclusion Criteria:

* Patients were diagnosed with nonmalignant breast disease
* Patients were offered neoadjuvant chemotherapy
* Patients had cognitive impairment
* Patients were physically unfit to be interviewed
* Patients were non-Mandarin or -Taiwanese

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Decisional conflict | 1 day before surgery
  Total score of decisional conflict scale
Knowledge | 1 day before surgery
  Total score on knowledge scale

SECONDARY OUTCOMES:
Decision regret | 4 weeks after surgery
  Total score of decision regret
Postsurgical depression | 4 weeks after surgery
  Total score of Hospital anxiety and depression scale (HADS)

CONTACTS AND LOCATIONS:
Overall Officials: Shared Decision Making Resource Center, Principal Investigator — Shuang Ho Hospital, Taipei Medical University
Locations (1):
- Shuang Ho Hospital, Taipei Medical University, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin SQ, Su CM, Wu HC, Chou YY, Yen YC, Tam KW. Effect of patient decision aids on decisional conflict and regret associated with breast cancer surgery: a randomized controlled trial. Breast Cancer. 2022 Sep;29(5):880-888. doi: 10.1007/s12282-022-01370-0. Epub 2022 May 19. PMID 35589905